CLINICAL TRIAL: NCT04737460
Title: Phase 1 Intrathecal Lumbar Administration of AAV9/CLN7 for Treatment of CLN7 Disease
Brief Title: Study for the Treatment for CLN7 Disease
Acronym: CLN7
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Benjamin Greenberg (Other)
Responsible Party: Sponsor-Investigator, Benjamin Greenberg, Professor of Neurology and Neurotherapeutics, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 2020-0640
Record Dates: First submitted 2021-01-15; First posted 2021-02-03 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: CLN7
Keywords: CLN7; Batten's Disease; AAV9/CLN7
MeSH Terms: conditions — Neuronal Ceroid-Lipofuscinoses

STUDY DESIGN:
Intervention Model Description: An initial low dose cohort followed by a subsequent a high dose cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AAV9/CLN7 (Experimental): AAV9/CLN7 is an intrathecally administered AAV9-based gene therapy vector that expresses the fully functional form of MFSD8 under the control of a synthetic promoter. AAV9/CLN7 is designed to achieve stable, potentially life-long expression of MFSD8 in non-dividing cells.
  The first participant will receive a low dose of 5X1014 vg, subsequent participants will receive a higher dose of 1x1015 vg of the AAV9/CLN7 agent.
  Interventions: Genetic: AAV9/CLN7

INTERVENTIONS:
Genetic: AAV9/CLN7 — Enrollees will receive gene therapy via a viral vector

SUMMARY:
This is a phase 1 open-label, single-administration of gene therapy agent AAV9/CLN7, administered intrathecally into the lumbar spinal cord region of pediatric patients with CLN7 Batten disease.

This study consists of a one-time injection of AAV9/CLN7. There are two Cohorts with a low dose and a high dose.

The primary objective for this clinical study is to evaluate safety. The secondary objective is to determine the efficacy of AAV9/CLN7.

The secondary outcome measures include motor, cognition and intelligence assessments.

The exploratory outcome measures include visual impairment assessment, cognitive evaluations, Brain magnetic resonance imaging (MRI), electroencephalogram (EEG), electrocardiogram (ECG) and echocardiogram (ECHO).

ELIGIBILITY:
Inclusion Criteria:

* 1-18 years of age
* Clinically symptomatic patients with diagnosis of CLN7 based upon molecular testing with homozygous or compound heterozygous and pathogenic mutations in MFSD8 gene with symptom onset before age 4
* Patients selected to be included in this study will have no more than moderate severity of the disease and will have to meet the following criteria; Not dependent on chronic invasive ventilatory support AND have either
* Expressive language sub test on Mullen and/or Vineland consistent with an age equivalent score of a 2 year 0 month old. This means they should have 20-50 words (all comprehensible) in their vocabulary and putting 2-3 words phrases in a sentence or,
* Patients can complete and obtain a score of 2-3 on GMFM sub domain E (Walking, Running & jumping) item 67 (ie With 2 hands held can walk 10 steps forward)
* Written informed consent provided by participant/parent/guardian and willingness to participate and comply with all the study related visits and procedures. Assent provided by children 10 -17 years old based on their ability to understand the risks and possible benefits, and the activities expected of them as participants.

Exclusion Criteria:

* Diagnosis of a second neurodegenerative disease or another genetic syndrome with a progressive course
* Hypersensitivity to any drugs used per procedural protocol
* Inability to tolerate anesthesia or study procedures
* Advanced stage disease defined by the use of chronic invasive ventilatory support (tracheostomy with ventilator dependence) and a non communicative status
* Concomitant illness that places patient at risk for gene transfer or gene transfer related procedures and immunosuppression
* Active, symptomatic viral infection (including but not limited to HIV or serology positive for Hepatitis B or C, or COVID-19) at the PI's discretion
* Bacterial infection requiring antibiotics within the 6 weeks prior to infusion
* New antiepileptic medications initiated within 90 days of infusion
* Status epilepticus within 30 days of infusion
* Generalized tonic-clonic seizure without returning to baseline within 24 hours of infusion
* Family is unwilling or unable to participate with required follow-up assessments
* Abnormal lab values that are clinically significant:

  * Platelet count < 100,000/mm3
  * Abnormal absolute neutrophil count (ANC) of < 1000/mm3
  * Persistent leukopenia or leukocytosis (Total white blood cell count < 3,000/mm or > 15,000/mm respectively)
  * Significant anemia (Hb <10 g/dL)
  * Abnormal prothrombin (PT) or partial thromboplastin time (PTT)
  * Abnormal liver function tests (>2 X ULN or > 2 X the baseline value at time of dosing)
  * Abnormal pancreatic enzymes (>2 X ULN or > 2 X the baseline value at time of dosing)
  * Renal impairment defined as urinary protein concentration greater than or equal to 0.2 g/L on 2 consecutive tests
  * Any other abnormal lab values that are clinically significant per PI's discretion
  * If labs are abnormal, these can be rechecked during the screening period. If labs normalize with or without intervention, patient can be enrolled at the discretion of PI.
* Contraindications for intrathecal administration of the product via lumbar puncture, such as bleeding disorders or other medical conditions (e.g., spina bifida or clotting abnormalities)
* Contraindications for MRI scans (including but not limited to cardiac pacemaker, metal in the eye, aneurysm clip in the brain, etc.)
* History of or current chemotherapy, radiotherapy, or other immunosuppression therapy within 30 days preceding screening (corticosteroid treatment may be permitted at the discretion of the PI)
* Receipt of any other investigational agent within the previous 3 months
* Positive Beta hCG pregnancy test (females of child bearing potential will have a pregnancy test on Day -1)
* Any other medical condition that puts the subject at increased risk of adverse events related to the investigational product or study-related procedures.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2021-05-04 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety measured by the incidence and severity of treatment related serious adverse events | Day 0 to 720
  Adverse event collection at scheduled visits. Lab results at scheduled visits. MRI Brain at Days 90, 180, 360, 720. Lumbar Puncture with Cerebral Spinal Fluid analysis at Days 90, 180, 360 and 720.

SECONDARY OUTCOMES:
Mean change in disease burden as measured by Clinical Global Impression Scale (CGI-S) | Baseline, 24 months
  Clinical Global Impression Scale (CGI) a 3 item observer rated scale that measures illness severity global improvement or change and therapeutic response.
  The CGI-S is rated on a 7-point scale, with the severity of illness scale using a range of responses from 1 (normal) through to 7 (amongst the most severely ill patients).
  Possible score ranges from 1-7, with highest score indicating the most severely ill patients.
Mean change in disease burden as measured by Early Clinical Drug Evaluation Program (ECDEU) | Baseline, 24 months
  The Early Clinical Drug Evaluation Program (ECDEU) version of the CGI asks that the clinician rate the patient relative to their past experience with other patients with the same diagnosis. Treatment response ratings should take account of both therapeutic efficacy and treatment-related adverse events and range from 0 (marked improvement and no side effects) to 4 (unchanged or worse and side effects outweigh the therapeutic effects).
  Possible scores range from 0-4, with lower score indicating more improvement.
Mean change in motor function as measured by 2- minute Walk Test | Baseline, 24 months
  Ataxia and Motor Function Assessments include a 2 - minute Walk test measuring endurance.
  The timed walk test will be completed by participants who can ambulate sufficiently. The Two Minute Walk Test (2MWT) measures the distance that an individual over age 3 can walk on a flat surface in a period of 2 minutes, and assesses endurance relative to the musculoskeletal, pulmonary, and cardiovascular systems.
Mean change in motor function as measured by 6- minute Walk Test | Baseline, 24 months
  Ataxia and Motor Function Assessments include a 6- minute Walk test measuring endurance.
  The Six Minute Walk Test (6MWT) measures endurance in a similar fashion using a time interval of 6 minutes and is a commonly used measure for evaluating outcomes in research for multiple different populations of children and adults.
Mean change in motor function as measured by Pediatric Balance scale | Baseline, 24 months
  The Pediatric Balance Scale is a 14-item test used to evaluate functional balance in children.
  It is an adapted version of the Berg Balance Scale.
  Possible score ranges from 0-56 , with highest score indicating better performance.
Mean change in motor function as measured by Gross Motor Function Measure-88 | Baseline, 24 months
  Gross Motor Function Measure is used to measure self initiated movement in ambulatory and non-ambulatory participants to evaluate changes in gross motor function over time.
  Possible score ranges from 0-3, with higher score indicating better motor function.
Mean change in Neuropsychological state as measured by Mullen scales. | Baseline, 24 months
  The Mullen Scales of Early Learning is a comprehensive Neuropsychological assessment of early language, motor and cognitive abilities. T scores are given for individual scales and the four cognitive scales (visual reception, fine motor, receptive language and expressive language) are combined to to yield a composite score of Early Learning. Each scale is comprised of interactive tasks with a scoring range for each item of zero to 5 points.
  Test ages are converted to normalized T-scores by using tables based on the child's age. T scores have the same meaning regardless of a child's age.
  Possible score ranges from 1-100 for percentile ranking, with higher score indicating higher performance.
Mean change in Neuropsychological state as measured by Vineland Adaptive Behavior Scales | Baseline, 24 months
  The Vineland Adaptive Behavior Scale is one of the most well-known and well-validated Neuropsychological measures of adaptive functioning. Four key domains will be rated including communication skills, daily living skills, social skills and motor skills. The combination of these makes up the overall Adaptive Behavior Composite (ABC). Scores are based on standard scores for the domains and age-equivalents meaning the scores are compared to that of others that are his or her age.
  The score is a percentile ranking in an individual's normative age group. The higher the percentage ranking indicates a better outcome on the scale.
  Possible score ranges from 1 -100 for percentile ranking, with higher score indicating higher performance.
Mean change of Quality of life as measured by Quality of Life Inventory - Disability questionnaire | Baseline, 24 months
  Quality of Life Inventory - Disability (QI-Disability) questionnaire measures quality of life with 32-item measures that includes - a child's social interactions, positive emotions, physical health, negative emotions, leisure skills, and independence. Scores are a 5-point Likert scale and then are transformed to a scale of 0 to 100.
  Possible scores range from 0-100, with higher scores indicating better quality of life.
Mean change of Quality of life as measured by Infant and Toddler Quality of Life Questionnaire (ITQOL) | Baseline, 24 months
  The ITQOL Short Form is a 47-item measure to assess physical and psychosocial functioning of children ages 2 months to 5 years. It contains 12 scales including physical functioning, growth and development, bodily pain, temperament and moods, general behavior, getting along, general health perceptions, parental impact-emotional, parental impact-time, family activities, family cohesion, and change in health. Scores are transformed to a scale of 0 to 100.
  Possible scores range from 0-100, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Greenberg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Children' Health, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No